CLINICAL TRIAL: NCT03043248
Title: TRK-700 Drug-Drug Interaction Study With Digoxin and Midazolam in Healthy Adults
Brief Title: TRK-700 Drug-Drug Interaction Study With Digoxin and Midazolam
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Toray Industries, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 700P1C03
Record Dates: First submitted 2017-02-02; First posted 2017-02-03 (Estimated); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Healthy
Keywords: TRK-700; PK; Digoxin; Midazolam; Drug-Drug interaction; P-glycoprotein; CYP3A4; MDR1; pharmacokinetics; multidrug resistance 1
MeSH Terms: interventions — Digoxin; Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort A (Experimental): TRK-700 + Digoxin
  Interventions: Drug: TRK-700; Drug: Digoxin
- Cohort B (Experimental): TRK-700 + Midazolam
  Interventions: Drug: TRK-700; Drug: Midazolam

INTERVENTIONS:
Drug: TRK-700 — repeated oral administration
Drug: Digoxin — single oral administration with/without TRK-700
  Arms: Cohort A
Drug: Midazolam — single oral administration with/without TRK-700
  Arms: Cohort B

SUMMARY:
This study comprises 2 cohorts, and in each cohort, the study will be conducted as an open-label add-on study.

The purpose of the study is to investigate the pharmacokinetics of each substrate in concomitant administration of a single dose of the P-glycoprotein substrate digoxin (Cohort A) or the CYP3A4 substrate midazolam (Cohort B) during repeated administration of TRK-700 in healthy adult males.

ELIGIBILITY:
Inclusion Criteria:

* Japanese healthy adult males.
* Subjects with a BMI of at least 18.0 and less than 30.0 at the screening examination and the examination at admission.

Exclusion Criteria:

* Subjects with significant concomitant or historical disease of the metabolism, liver, kidneys, blood, lungs, heart, digestive organs, urinary organs, or nerves, or psychiatric diseases, accompanied by clinical symptoms or with other clinically significant disease, who are unsuitable for participation in this study, in the opinion of the investigators.
* Subjects who are found by the investigators to have significant clinical abnormality at the screening examination, the examination at admission, or the examination at the day of first administration of Digoxin or Midazolam.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2017-02-06 (Actual); Primary Completion 2017-05-13 (Actual); Study Completion 2017-05-21 (Actual)

PRIMARY OUTCOMES:
Area under the plasma drug concentration - time curve from administration to the last available concentration measurement of Digoxin and Midazolam(AUClast) | Cohort A: up to 72 hours, Cohort B: up to 48 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Tokyo, Tokyo, Japan